CLINICAL TRIAL: NCT00244673
Title: Diphteria-tetanus-pertussis (DTP) Vaccination and Child Survival: Randomized Study of Not Providing DTP Vaccination Together With or After Measles Vaccination
Brief Title: Randomized Study of Not Giving Diphteria-tetanus-pertussis Vaccination With or After Measles Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: Aarhus University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CVEK2005-7041-45-DTPMV; CVEK2005-7041-45
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Mortality; Hospitalization; Adverse Events
Keywords: Vaccination; DTP; Child mortality; Sex; Non-specific effects
MeSH Terms: conditions — Coitus

INTERVENTIONS:
Biological: DTP3/4+OPV+MV versus OPV+MV or DTP4+OPV4 versus OPV4 — Trial of not providing 3. and/or 4. DTP together with or after MV at 9 to 18 month of age.

SUMMARY:
In non-randomized studies, routine childhood vaccinations have been observed to have non-targeted effects. Difteria-tetanus-pertussis (DTP) vaccine provided with or after measles vaccine (MV) is associated with increased mortality in areas with herd immunity to pertussis.

We will examine in a randomised study of 6000 children the effect of not administering DTP simultaneously with or after MV on overall child mortality, hospitalization rates, and the immunological responses after vaccination. We will also examine potential sex-differential effects in the outcomes and interactions with other vaccines, other health interventions and season.

DETAILED DESCRIPTION:
Background: Infectious diseases are the main cause of high child mortality in Africa. In several non-randomised studies, routine childhood vaccinations have been observed to have non-targeted effects. Live vaccines like measles vaccine (MV) seem to protect against overall mortality, whereas killed vaccines, like DTP, may have no beneficial effects, especially for girls. DTP provided with or after MV may be associated with increased mortality. The mechanisms behind these effects are unknown.

Hypothesis: Not providing DTP together with or after MV is associated with a 35 % reduction in overall mortality and 23% reduction in hospitalizations.

Objectives: To examine in a randomised study of 6000 children the effect of not administering DTP simultaneously with or after MV on

1. Overall child mortality
2. Hospitalization rates and major causes of hospitalization
3. The immunological profile after vaccination
4. Sex-differences in the above mentioned outcomes

Methods:

Surveillance system: BHP's demographic surveillance system in Bissau covers 6 districts with a population of 90,000; 3,500 children are born each year.

Hospitalizations: There is only one pediatric ward in Bissau and all hospitalizations are identified in the BHP register.

Vaccinations: Vaccinations are provided and registered at the 3 health centres in the study area.

Intervention: In this study 6000 children are randomised as they come to receive DTP3 or DTP booster with or after measles vaccination (MV) at the local health centres. Children will be randomised to DTP3+OPV3 and MV versus OPV3 and MV or DTP4+OPV4 versus OPV4 (booster doses).

Follow-up: The children will be followed until 4 years of age or end of study.

1. Adverse effects: In the first month after vaccination, 1000 children will be visited daily for three days and then weekly to register morbidity and consultations.
2. Hospitalizations: The children will be followed at the pediatric ward.
3. Mortality: Children will be followed by the routine surveillance system. Furthermore, all children will be visited yearly and finally when they reach four years of age. When a death is detected, a physician will conduct a verbal autopsy.

Sample size: With a total of 7500 person-years of follow-up, we will be able to document a 35% reduction in mortality and a 23% reduction in hospitalizations. A subgroup of children will be examined for possible differences in immunological profile after vaccination.

Ethical considerations: Herd immunity to pertussis should not be affected as, due to the intervention, more children is vaccinated.

ELIGIBILITY:
Inclusion Criteria:

1. The child should be missing DTP3 or DTP4
2. The child should have received DTP2
3. The child should have received MV already or receive MV on the day of enrolment

Exclusion Criteria:

Normally applied contraindications for receiving vaccinations, including high fever

Ages: 9 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6534 (Actual)
Dates: Start 2005-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Mortality till 4 years of age | June 2011
Hospitalisations till 4 years of age | June 2011
Adverse events 1 month after intervention | December 2008

SECONDARY OUTCOMES:
Immunological responses | July 2008
Morbidity | June 2011

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, DMSc, Principal Investigator — Bandim Health Project
Locations (1):
- Bandim Health Project, Apartado 861, Bissau, Guinea-Bissau